CLINICAL TRIAL: NCT04104035
Title: A Comparative Study of Leukemic Stem Cells in Patients With BCR-ABL-positive Hematopoiesis and Chronic Myeloid Leukemia Patients With BCR-ABL Activity Inhibition Under Tyrosine Kinase Inhibitor Treatment
Brief Title: Leukemic Stem Cell Detection for Chronic Myeloid Leukemia Patients With Major Molecular Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Osman Ilhan, Prof., Ankara University
Other Study IDs: CML-BCR-ABL-TKI
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; BCR-ABL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples from 30 patients and bone marrow aspiration samples from 20 patients will be collected for each group. A total of 100 patients will be included in the study. The number of bone marrow aspiration samples is limited to 20 patients for each group, as this method is more invasive with a higher rate of complications. Peripheral blood samples will be collected simultaneously in patients in whom bone marrow samples are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BCR-ABL-positive hematopoiesis: Patients with BCR-ABL-positive hematopoiesis (newly diagnosed CML patients, CML patients with leukocytosis, CML patients without a hematological and/or cytogenetic and/or molecular response, CML patients whose BCR-ABL status becomes negative and then positive) will be included.
- BCR-ABL activity inhibition under TKI: Patients with CML with BCR-ABL activity inhibition under TKI therapy (patients with MMR and/or deeper response) will be included.

SUMMARY:
Multi-Center, national, non-drug, prospective cohort study Target patient number is 100 The amount of CD45+/CD34+/CD38-/CD26+ levels of chronic myeloid leukemia (CML) stem cells in CML patients with and without BCR-ABL hematopoiesis will be compared.

There will be 2 arms;

1. Patients with BCR-ABL-positive hematopoiesis
2. CML patients with BCR-ABL activity inhibition under tyrosine kinase inhibitor (TKI) therapy

DETAILED DESCRIPTION:
In the present study, its aimed to compare the amount of CD45+/CD34+/CD38-/CD26+ levels of CML stem cells in CML patients with and without BCR-ABL hematopoiesis. Therefore, the amount of CD45+/CD34+/CD38-/CD26+ levels of CML stem cells in CML patients will be analyzed using bone marrow and peripheral blood samples and whether leukemic stem cells are present in the bone marrow and at what amount, if present, although these cells are cleared from the peripheral blood, will be investigated. Additionally this study would pave the way for further cellular treatment strategies against CML stem cells, being the pioneer of development of curative treatments in CML. Until now, TKI discontinuation studies have failed in patients with long-term BCR-ABL negativity. There is a chance for cure in patients in whom the BCR-ABL status becomes negative with chimeric antigen receptor (CAR) T-cell treatment modalities which target leukemic stem cells. Also, monoclonal antibodies and/or cellular treatments targeting leukemic stem cells are the main treatment strategy is to reduce the CML treatment-related cost. In the international platform, the accurate definition of leukemic stem cell in CML and development of targeted cellular treatments have been also paid a great attention with a given priority for patent application. The primary objective of the present study is to accurately detect leukemic stem cells in CML and to estimate the threshold value for the prediction of recurrence or cure.

To the best of investigators knowledge, there is a very limited number of studies in the literature and there is no study available comparing leukemic stem cells (CD45+/CD34+/CD38-/CD26+) in patients with BCR-ABL-positive hematopoiesis and CML patients with BCR-ABL activity inhibition under TKI therapy in Turkey. Therefore,for the first time, it is planned to evaluate the prognostic value of the amount of leukemic stem cells in CML and to tailor individual treatment options.

Newly diagnosed CML patients or patients with a previous diagnosis under follow-up with or without TKIs will be included in this study. The patients will be divided into two groups as follows:

Group 1: Patients with BCR-ABL-positive hematopoiesis (newly diagnosed CML patients, CML patients with leukocytosis, CML patients without a hematological and/or cytogenetic and/or molecular response, CML patients whose BCR-ABL status becomes negative and then positive) will be included.

Group 2: Patients with CML with BCR-ABL activity inhibition under TKI therapy (patients with major molecular response (MMR) and/or deeper response) will be included.

Peripheral blood samples from 30 patients and bone marrow aspiration samples from 20 patients will be collected for each group. A total of 100 patients will be included in the study. The number of bone marrow aspiration samples is limited to 20 patients for each group, as this method is more invasive with a higher rate of complications. Peripheral blood samples will be collected simultaneously in patients in whom bone marrow samples are collected. For an accurate examination, the bone marrow samples and the peripheral blood samples will be concomitantly analyzed for each individual patient. The presence and amount of CD45+/CD34+/CD38-/CD26+ leukemic stem cells will be analyzed using multicolor flow cytometry at Ankara University, Faculty of Medicine, Ibni Sina Hospital, Hematology Lab. The peripheral blood and bone marrow samples obtained at Hacettepe University and Ege University will be transferred to Ankara University, Faculty of Medicine, Ibni Sina Hospital, Hematology Lab in accordance with the codes of the Biological Material Transfer Agreement. As bone marrow aspiration and BCR-ABL molecular testing are routinely used in the diagnosis and follow-up of CML patients, these interventions pose no additional burden for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed CML patients or patients with a previous diagnosis under follow-up with TKIs

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed CML patients or patients with a previous diagnosis under follow-up with or without TKIs will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Detection of CML leukemic stem cells in both peripheral blood and bone marrow of CML patients | 1 day
  To detect the leukemic stem cells using an accurate, simple, and accessible tool in CML patients

SECONDARY OUTCOMES:
Detection of CML leukemic stem cell in bone marrow of patients in whom BCR-ABL is negative in peripheral blood with TKIs | 1 day
  The data obtained from these patients may identify the dynamics of CML leukemic stem cell in bone marrow and role of stem cell response under TKIs that can more accurately predict the success of discontinuation of TKIs.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Ilhan, Prof, Principal Investigator — Ankara University Medical Faculty Department of Hematology
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No